CLINICAL TRIAL: NCT00000306
Title: Dextroamphetamine as an Adjunct in Cocaine/Opiate Dependent Patients
Brief Title: Dextroamphetamine as Adjunct in Cocaine/Opiate Dependent Patients - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09262-3; P50-09262-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Dextroamphetamine

INTERVENTIONS:
Drug: Dextroamphetamine

SUMMARY:
The purpose of this study is to evaluate dextroamphetamine sulfate (sustained release) as an adjunct in concurrent cocaine and opiate dependent patients.

DETAILED DESCRIPTION:
This 27-week double-blind, placebo controlled treatment is designed to evaluate dextroamphetamine sulfate (sustained release) as an adjunct in concurrent cocaine and opiate dependent patients. All subjects will receive methadone. For the treatment of cocaine dependence, subjects will receive one of 2 doses of dextroamphetamine (15 or 30mg) or placebo. After 4 weeks of treatment the dose level of dextroamphetamine is doubled (30 or 60mg). This dose is maintained for 20 weeks; during which subjects attend twice weekly visits to the clinic and receive weekly cognitive behavioral therapy. Follow up evaluations will be conducted out to 3 months post treatment. Subjects will be assisted in transferring to Houston area methadone clinics to maintain treatment for opiate dependence following treatment completion.

ELIGIBILITY:
Inclusion Criteria- Subject must:

* Exhibit cocaine and opiate dependence through a DSM-IV diagnosis as determined by SCID.
* Be between 18 and 45 years old
* Women must agree to use contraception
* Have an EKG that has been confirmed by a cardiologist
* Give a cocaine positive urine during screening - Present with evidence of opiate withdrawal

Exclusion Criteria- Subject must not:

• Have a serious medical illness including, but not limited to the following: Hypertension Significant heart disease Clinically significant cardiovascular abnormality Angina Hepatic, renal, or gastrointestinal disorders that could result in an altered metabolism or excretion of study agent

* Have any Axis I disorder that is not related to drug use
* Have current dependence on any psychoactive disorder other than nicotine
* Be on probation or parole for reasons other than those related to drug charges (ASI)
* Be pregnant or lactating
* Have been in any outside treatment in 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 1994-09; Study Completion 2001-09

PRIMARY OUTCOMES:
Craving
Drug use
Medication compliance
Retention
Addiction severity
Mood indicators
Psychiatric interview

SECONDARY OUTCOMES:
Effectiveness measures including psycho-social variables, side effects, and self-reported measures.

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States